CLINICAL TRIAL: NCT00483704
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group Multiple Attacks Study to Compare the Efficacy and Safety of Oral MK-0974 With Placebo for the Acute Treatment of Migraine With or Without Aura
Brief Title: Multiple Attacks Study to Compare the Efficacy and Safety of MK-0974 With Placebo for Acute Migraine (MK-0974-031)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-031; MK-0974-031 (Other: Merck Protocol Number); 2007_546 (Other: Telerx ID Number)
Record Dates: First submitted 2007-05-15; First posted 2007-06-07 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Migraines
Keywords: multiple attacks of moderate to severe migraine headaches
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telcagepant 140 mg (Experimental): Telcagepant 140 mg, oral, tablet, across 4 migraine attacks. For migraine attack 1 only, if no headache relief is obtained after 2 hours post dose, or if the migraine recurs after 2 hours of the initial treatment, participants may receive an optional second dose of telcagepant 140 mg or placebo.
  Interventions: Drug: Telcagepant 140 mg
- Telcagepant 280 mg (Experimental): Telcagepant 280 mg, oral, tablet, across 4 migraine attacks. For migraine attack 1 only, if no headache relief is obtained after 2 hours post dose, or if the migraine recurs after 2 hours of the initial treatment, participants may receive an optional second dose of telcagepant 280 mg or placebo.
  Interventions: Drug: Talcagepant 280 mg
- Control Group 1 (Placebo Comparator): Placebo, oral, tablet, across 3 migraine attacks (1st, 2nd, and 4th). Telcagepant 140 mg will be administered for the 3rd migraine attack. Participants will receive placebo for the optional second dose. For migraine attacks 2, 3, and 4, no study medication will be provided as an optional second dose.
  Interventions: Drug: Telcagepant 140 mg; Drug: Placebo
- Control Group 2 (Placebo Comparator): Placebo, oral, tablet, across 3 migraine attacks (1st, 2nd, and 3rd). Telcagepant 140 mg will be administered for the 4th migraine attack. Participants will receive placebo for the optional second dose. For migraine attacks 2, 3, and 4, no study medication will be provided as an optional second dose.
  Interventions: Drug: Telcagepant 140 mg; Drug: Placebo

INTERVENTIONS:
Drug: Telcagepant 140 mg — Telcagepant 140 mg tablets
  Arms: Control Group 1; Control Group 2; Telcagepant 140 mg
Drug: Talcagepant 280 mg — Telcagepant 280 mg tablets
  Arms: Telcagepant 280 mg
Drug: Placebo — Placebo tablets
  Arms: Control Group 1; Control Group 2

SUMMARY:
The purpose of the study is to assess the safety and efficacy of telcagepant (MK-0974) in acute treatment of multiple migraine attacks with or without aura. Primary hypotheses of this study are that telcagepant is superior to placebo, as measured by the proportion of participants who have pain freedom, pain relief, pain freedom consistency, pain relief consistency, and absence of photophobia, phonophobia, and nausea at 2 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* History of migraines within the past year
* 1 to 8 moderate or severe migraine attacks per month in the past 2 months that lasted between 4 to 72 hours if untreated
* Use acceptable contraception throughout the study
* Able to complete the study questionnaire(s) and paper diary
* Limit consumption of grapefruit juice to no more than one 8 ounce glass a day

Exclusion Criteria:

* Pregnant or breast-feeding or is expecting to become pregnant during the study
* Difficulty distinguishing his/her migraine attacks from tension or interval headaches
* A history of mostly mild migraine attacks or migraines that usually resolve spontaneously in less than 2 hours
* More than 15 headache-days per month or has taken medication for acute headache on more than 10 days a month in the past 3 months
* Greater than 50 years old at the age of migraine onset
* Previously taken telcagepant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1935 (Actual)
Dates: Start 2008-08-14 (Actual); Primary Completion 2009-03-25 (Actual); Study Completion 2009-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ho AP, Dahlof CG, Silberstein SD, Saper JR, Ashina M, Kost JT, Froman S, Leibensperger H, Lines CR, Ho TW. Randomized, controlled trial of telcagepant over four migraine attacks. Cephalalgia. 2010 Dec;30(12):1443-57. doi: 10.1177/0333102410370878. Epub 2010 Jun 8. PMID 20974601
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-031&kw=0974-031&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Telcagepant 140 mg: Telcagepant 140 mg, oral, across 4 migraine attacks. For migraine attack 1 only, if no headache relief is obtained after 2 hours post dose, or if the migraine recurs after 2 hours of the initial treatment, participants may receive an optional second dose of telcagepant 140 mg or placebo.
- Telcagepant 280 mg: Telcagepant 280 mg, oral, across 4 migraine attacks. For migraine attack 1 only, if no headache relief is obtained after 2 hours post dose, or if the migraine recurs after 2 hours of the initial treatment, participants may receive an optional second dose of telcagepant 280 mg or placebo.
- Placebo: The placebo group is comprised of Control Group 1 and Control Group 2. Control Group 1 receives placebo across 3 migraine attacks (1st, 2nd, and 4th) and telcagepant 140 mg for the 3rd migraine attack. Control Group 2 receives placebo across 3 migraine attacks (1st, 2nd, and 3rd) and telcagepant 140 mg for the 4th migraine attack. For both groups for migraine attacks 2, 3, and 4, no study medication will be provided as an optional second dose.
Period: Randomization
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Started | 644 | 645 | 646
Completed | 573 | 549 | 555
Not Completed | 71 | 96 | 91
Not completed — Withdrawal by Subject | 19 | 28 | 18
Not completed — Protocol Violation | 14 | 25 | 22
Not completed — Lost to Follow-up | 14 | 14 | 19
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 0
Not completed — Progressive disease | 0 | 0 | 1
Not completed — Lack of qualifying migraines | 21 | 25 | 31
Period: Treatment
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Started | 573 | 549 | 555
Completed | 444 | 420 | 399
Not Completed | 129 | 129 | 156
Not completed — Lack of qualifying migraines | 101 | 99 | 116
Not completed — Adverse Event | 3 | 5 | 4
Not completed — Withdrawal by Subject | 16 | 12 | 21
Not completed — Protocol Violation | 6 | 3 | 5
Not completed — Lost to Follow-up | 2 | 7 | 5
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo | Total
Number analyzed (Participants) | 644 | 645 | 646 | 1935
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (11.7) | 42.6 (11.8) | 41.9 (11.7) | 42.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542 | 549 | 540 | 1631
  Male | 102 | 96 | 106 | 304

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pain Freedom at 2 Hours Post-dose (First Migraine Attack)
Description: Pain Freedom (PF) at 2 hours post-dose (first migraine attack), with pain freedom defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 0 at 2 hours post-dose. Headache severity was subjectively rated by the participant at predefined time points on a scale of Grade 0 to Grade 3: Grade 0 - No pain; Grade 1 - Mild pain; Grade 2 - Moderate Pain; and Grade 3 - Severe Pain.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: The full-analysis set (FAS) included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline pain score or post-dose data through 2 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 556 | 534 | 539
Percentage of participants | 21.9 | 25.1 | 10.2
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.80 to 3.58] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.03, 95% CI 2-sided [2.15 to 4.27] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

2. Primary Outcome: Percentage of Participants Reporting Pain Relief at 2 Hours Post-dose (First Migraine Attack)
Description: Pain Relief (PR) at 2 hours post-dose (first migraine attack), with pain relief defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 1/0 at 2 hours post-dose. Headache severity was subjectively rated by the participant at predefined time points on a scale of Grade 0 to Grade 3: Grade 0 - No pain; Grade 1 - Mild pain; Grade 2 - Moderate Pain; and Grade 3 - Severe Pain.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline pain score or post-dose data through 2 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 556 | 534 | 539
Percentage of participants | 58.6 | 56.7 | 33.4
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.03, 95% CI 2-sided [2.35 to 3.90] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.80, 95% CI 2-sided [2.17 to 3.61] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

3. Primary Outcome: Percentage of Participants Reporting Pain Freedom Consistency at 2 Hours Post-dose
Description: Pain Freedom Consistency (PFC) at 2 hours post-dose, defined as having achieved PF at 2 hours post-dose on at least 3 treated migraine attacks. Note that for the control groups, a positive PF response arising from the administration of the 1 talcagepant treated migraine attack will count as one of the 3 positive PF responses needed to fulfill the criteria for PFC.
Time Frame: 2 hours post-dose (up to 6 months)
Population: The modified FAS (MFAS) Population consisted of all participants who experienced at least either 2 failures or 3 successes, regardless of whether or not they had data for 4 migraine attacks, and recorded baseline severity for at least 1 of the treated migraine attacks.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 493 | 468 | 485
Percentage of participants | 9.3 | 14.1 | 2.7
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.85, 95% CI 2-sided [2.05 to 7.23] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 6.18, 95% CI 2-sided [3.36 to 11.39] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

4. Primary Outcome: Percentage of Participants Reporting Pain Relief Consistency at 2 Hours Post-dose
Description: Pain Relief Consistency (PRC) at 2 hours post-dose, defined as having achieved PR at 2 hours post-dose on at least 3 treated migraine attacks. Note that for the control groups, a positive PR response arising from the administration of the 1 telcagepant treated migraine attack will count as one of the 3 positive PR responses needed to fulfill the criteria for PRC.
Time Frame: 2 hours post-dose (up to 6 months)
Population: The MFAS Population was defined as all participants who experienced at least either 2 failures or 3 successes, regardless of whether or not they had data for 4 migraine attacks, and recorded baseline severity for at least 1 of the treated migraine attacks.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 469 | 440 | 452
Percentage of participants | 41.8 | 46.8 | 22.3
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.96 to 3.51] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.23, 95% CI 2-sided [2.41 to 4.34] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

5. Primary Outcome: Percentage of Participants Reporting Absence of Photophobia at 2 Hours Post-dose (First Migraine Attack)
Description: The participant recorded whether photophobia (sensitivity to light) was present or absent at each of the predefined time points.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose measurement for photophobia severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline photophobia score or post-dose data through 2 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 554 | 534 | 539
Percentage of participants | 52.3 | 52.4 | 40.6
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.30 to 2.11] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.31 to 2.14] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

6. Primary Outcome: Percentage of Participants Reporting Absence of Phonophobia at 2 Hours Post-dose (First Migraine Attack)
Description: The participant recorded whether phonophobia (sensitivity to sound) was present or absent at each of the predefined time points.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose phonophobia measurement prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline phonophobia score or post-dose data through 2 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 555 | 534 | 537
Percentage of participants | 61.4 | 59.4 | 48.6
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.36 to 2.22] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.26 to 2.06] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

7. Primary Outcome: Percentage of Participants Reporting Absence of Nausea 2 Hours Post-dose (First Migraine Attack)
Description: The participant recorded whether nausea was present or absent at each of the predefined time points.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose measurement for nausea severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline nausea score or post-dose data through 2 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 553 | 534 | 538
Percentage of participants | 72.9 | 71.7 | 62.8
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.28 to 2.17] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.21 to 2.04] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

8. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE) Within 48 Hours Post-dose (First Migraine Attack)
Description: AEs were reported following treatment for the first migraine attack using a 48-hour post-dose window. AEs displayed are those reported by at least 4 participants in one or more treatment groups.
Time Frame: Up to 48 hours post-dose for the first migraine attack (up to 6 months)
Population: The All-Patients-as-Treated (APaT) Population consisted of all participants who received at least 1 dose of study medication and were included in the treatment group according to the medication actually received. If a participant took an unassigned study medication for the first migraine attack, they were included in that treatment group.
Measure: Number; unit: Participants
Groups:
- Telcagepant 140 mg: Participants who received at least one dose of telcagepant 140 mg.
- Telcagepant 280 mg: Participants who received at least one dose of telcagepant 280 mg.
- Placebo: Participants who received at least one dose of placebo.
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 575 | 538 | 564
Participants | 179 | 167 | 157

9. Primary Outcome: Number of Participants Discontinuing Study Medication Due to an AE
Description: Participants discontinuing study medication due to an AE were reported for all migraine attacks.
Time Frame: Up to the 4th dose of study medication (up to 6 months)
Population: The APaT Population consisted of all participants who received at least 1 dose of study medication and were included in the treatment group according to the medication actually received. If a participant took an unassigned study medication, they were included in that treatment group.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 573 | 543 | 561
Participants | 3 | 5 | 4

10. Secondary Outcome: Percentage of Participants Reporting Sustained Pain Freedom From 2 to 24 Hours Post-dose (First Migraine Attack)
Description: Sustained Pain Freedom (SPF) from 2 to 24 hours after study medication administration. SPF from 2 to 24 hours post-dose is defined as PF at 2 hours, with no administration of either rescue medication or the optional second dose and with no occurrence thereafter of a mild/moderate/severe headache during the 2 to 24 hours after dosing with the study medication.
Time Frame: From 2 to 24 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population was participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hr. time point. Participants were excluded from this analysis for not having a baseline pain score, post-dose data through 24 hrs, or a recurrence question.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 553 | 529 | 537
Percentage of participants | 15.6 | 19.1 | 6.5
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.78 to 4.07] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.45, 95% CI 2-sided [2.30 to 5.19] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

11. Secondary Outcome: Percentage of Participants Reporting Sustained Pain Freedom From 2 to 48 Hours Post-dose (First Migraine Attack)
Description: Sustained Pain Freedom (SPF) from 2 to 48 hours post-dose after study medication administration. SPF from 2 to 48 hours post-dose is defined as PF at 2 hours, with no administration of either rescue medication or the optional second dose and with no occurrence thereafter of a mild/moderate/severe headache during the 2 to 48 hours after dosing with the study medication.
Time Frame: From 2 to 48 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population was participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hr. time point. Participants were excluded from this analysis for not having a baseline pain score, post-dose data through 48 hrs, or a recurrence question.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 552 | 526 | 536
Percentage of participants | 13.4 | 17.9 | 6.2
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.56 to 3.69] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.37, 95% CI 2-sided [2.22 to 5.12] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

12. Secondary Outcome: Percentage of Participants Reporting Total Migraine Freedom at 2 Hours Post-dose (First Migraine Attack)
Description: TMF 2 hours post-dose, which is defined as TMF at 2 hours post-dose, with no administration of either rescue medication or the optional second dose and with no occurrence thereafter of a mild/moderate/severe headache and no reported occurrence of photophobia, phonophobia, nausea, or vomiting during the 2 hours after dosing with the study medication.
Time Frame: 2 hours post-dose for the first migraine attack (up to 6 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 556 | 534 | 539
Percentage of participants | 19.4 | 22.3 | 9.5
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.65 to 3.38] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.97 to 4.01] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

13. Secondary Outcome: Percentage of Participants Reporting Total Migraine Freedom From 2 to 24 Hours Post-dose (First Migraine Attack)
Description: TMF from 2 to 24 hours post-dose, which is defined as TMF at 2 hours post-dose, with no administration of either rescue medication or the optional second dose and with no occurrence thereafter of a mild/moderate/severe headache and no reported occurrence of photophobia, phonophobia, nausea, or vomiting during the 2 to 24 hours after dosing with the study medication.
Time Frame: From 2 to 24 hours post-dose for the first migraine attack (up to 6 months)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline pain score or post-dose data through 24 hours.
Measure: Number; unit: Percentage of participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 553 | 531 | 537
Percentage of participants | 13.7 | 17.1 | 6.5
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.52 to 3.54] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 280 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 3.02, 95% CI 2-sided [2.00 to 4.56] — An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison

ADVERSE EVENTS:
Time Frame: Up to 14 days post-dose (up to 6 1/2 months)
Description: The APaT Population consisted of all participants who received at least 1 dose of study medication and were included in the treatment group according to the medication actually received. If a participant took an unassigned study medication, they were included in that treatment group.
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/573 | 8/543 | 4/561
Other Adverse Events (participants affected / at risk) | 166/573 | 144/543 | 138/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telcagepant 140 mg (N=573) | Telcagepant 280 mg (N=543) | Placebo (N=561)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telcagepant 140 mg (N=573) | Telcagepant 280 mg (N=543) | Placebo (N=561)
Dry mouth (Gastrointestinal disorders) | 61 (98) | 42 (82) | 53 (105)
Nausea (Gastrointestinal disorders) | 44 (59) | 47 (65) | 37 (54)
Fatigue (General disorders) | 48 (64) | 34 (43) | 27 (44)
Dizziness (Nervous system disorders) | 36 (54) | 40 (57) | 40 (59)
Somnolence (Nervous system disorders) | 36 (54) | 32 (49) | 15 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.